CLINICAL TRIAL: NCT06242834
Title: Phase II, Single Arm, Open Label, Study of the Combination of Pembrolizumab and Tazemetostat to Overcome Immune Tolerance Following ASCT or CAR T-Cell Therapy in Patients With Aggressive B-Cell Non-Hodgkin's Lymphoma
Brief Title: Pembrolizumab and Tazemetostat to Overcome Immune Tolerance Following ASCT or CAR T-cell Therapy in Patients With Aggressive B-Cell Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 23H05; NCI-2024-00285 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00220351; NU 23H05 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Specimen Handling; pembrolizumab; Magnetic Resonance Spectroscopy; tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, tazemetostat) (Experimental): Starting on day 14 after standard of care ASCT or CAR-T cell treatment patients receive pembrolizumab IV on day 1 of each cycle. Starting cycle 2, patients receive tazemetostat PO BID on days 1-21 of each cycle. Cycles repeat every 21 days for 12 months in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography during screening, CT scan, PET scan, and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Drug: Tazemetostat

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; Keytruda; Lambrolizumab; MK-3475; Pembrolizumab Biosimilar BCD-201; SCH 900475
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Tazemetostat — Given PO
  Other Names: E7438; EPZ-6438; EPZ6438

SUMMARY:
This phase II trial tests how well pembrolizumab and tazemetostat work to treat patients who have received autologous stem cell transplantation (ASCT) or chimeric antigen receptor (CAR) T cell therapy for aggressive non hodgkins lymphoma. A monoclonal antibody, such as pembrolizumab, is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Tazemetostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab and tazemetostat may work better to treat patients who have received ASCT or CAR-T cell therapy for aggressive non hodgkins lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the event-free survival (EFS) for the combination of pembrolizumab and tazemetostat as maintenance for 12 months in patients with aggressive B-cell Non- Hodgkin's Lymphoma following ASCT or CAR T-cell therapy.

SECONDARY OBJECTIVES:

I. To assess the progression-free survival (PFS) for the combination of pembrolizumab and tazemetostat as maintenance for 12 months in patients with aggressive B-cell Non-Hodgkin's Lymphoma following ASCT or CAR T-cell therapy.

II. To assess the overall survival (OS) for the combination of pembrolizumab and tazemetostat as maintenance for 12 months in patients with aggressive B-cell Non-Hodgkin's Lymphoma following ASCT or CAR T-cell therapy.

III. To evaluate the safety and toxicity of the combination of pembrolizumab and tazemetostat as maintenance therapy for 12 months following ASCT or CAR T cell therapy.

IV. To determine the objective response rate (ORR), complete response (CR) rate and partial response (PR) rate in patients receiving CAR T-cell therapy during maintenance phase (as assessed by Lugano Criteria).

EXPLORATORY OBJECTIVES:

I. To assess the change in immune cell subsets and cytokines, measured by flow and proteomics, with pembrolizumab alone and in combination with tazemetostat.

II. To determine survival outcomes (event free survival [EFS], PFS and OS) by type of treatment and line of therapy (ASCT, CAR T-cell therapy in second and third line).

OUTLINE:

Starting on day 14 after standard of care ASCT or CAR-T cell treatment patients receive pembrolizumab intravenously (IV) on day 1 of each cycle. Starting cycle 2, patients receive tazemetostat orally (PO) twice daily(BID) on days 1-21 of each cycle. Cycles repeat every 21 days for 12 months in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography during screening, computed tomography (CT) scan, positron emission tomography (PET) scan, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up within 90 days and periodically for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histo-pathologically confirmed aggressive B-cell NHL intended for or currently undergoing standard of care ASCT or CAR T-cell therapy.

  * Note: Patients should have met the Food and Drug Administration (FDA) approved indications for the respective CAR T cell construct being used. Standard of care/FDA approved CAR-Ts for this population include axicabtagene ciloleucel, tisagenlecleucel or lisocabtagene maraleucel, any of which may have been used for this patients and is provider dependent. Out of specification products of these respective CAR Ts may also be utilized if intended for FDA approved indication by way of expanded access if the provider feels that the product offers similar efficacy and safety as compared to commercial product per guidance provided by manufacturer. For the purpose of this study, aggressive B-cell NHL histologies should conform to the label indications for the respective CAR-T being utilized. Accordingly, CAR-T eligible histologies include the following groups according to the 2016 revision of the World Health Organization (WHO) classification of lymphoid neoplasms High-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements
  * High-grade B-cell lymphoma, Not Otherwise Specified (NOS)
  * Diffuse large B-cell lymphoma (DLBCL), NOS
  * Diffuse large B-cell lymphoma (DLBCL), NOS; Germinal center B-cell type** [Refer note below]
  * Diffuse large B-cell lymphoma (DLBCL), NOS; Non-germinal center B cell type** [Refer note below]
  * Large B-cell lymphoma with IRF4 rearrangement (subtype of DLCBL)
  * T-cell/histiocyte-rich large B-cell lymphoma (subtype of DLCBL)
  * Primary cutaneous DLBCL, leg type (subtype of DLCBL)
  * Epstein Barr Virus (EBV)+ DLBCL, NOS (subtype of DLCBL)
  * DLBCL associated with chronic inflammation (subtype of DLCBL)
  * Primary mediastinal (thymic) large B-cell lymphoma
  * Intravascular large B-cell lymphoma (subtype of DLCBL)
  * Transformed indolent B-cell lymphoma; composite lymphomas with aggressive B-cell NHL as outlined above and indolent lymphomas are also allowable if felt to represent transformation.

    * NOTE: * Cell of origin will be determined by Hans criteria (immuno histochemistry). We have therefore updated criteria to indicate non-germinal center B-cell type to reflect this (rather than activated B-cell [ABC] subtype which implies use of molecular testing)
* For CAR T-cell therapy, patients must have metabolically active disease on PET/CT prior to therapy; For ASCT therapy, patients must be in complete remission
* Patients must be age ≥ 18 years on the day of signing informed consent
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must have a life expectancy of greater than 12 weeks
* Absolute neutrophil count (ANC)* ≥ 500/μL neutrophil count prior to either admission for ASCT or CAR T-cell apheresis Note: * Use of growth factor is allowable if deemed clinically appropriate by the treating physician up to the day prior to LDC/conditioning chemotherapy (i.e. if felt to be disease related) Patients must meet the parameter at screening if intended for ASCT or CAR-T treatment but have not yet received the cellular therapeutic. For patients enrolled after receiving ASCT or CAR T-cell therapy, patients will be eligible if they meet the criteria on day 1 of either conditioning chemotherapy (ASCT) or lymphodepleting chemotherapy (LDC) (CAR-T)
* Platelets (PLT) ≥ 50,000/μL within 14 days prior to either admission for ASCT or CAR T-cell apheresis, unless deemed to be related to disease (transfusion not permitted within 7 days) Minimum platelet count requirement in those with bone marrow involvement will be ≥ 25,000 Patients must meet the parameter at screening if intended for ASCT or CAR-T treatment but have not yet received the cellular therapeutic. For patients enrolled after receiving ASCT or CAR T-cell therapy, patients will be eligible if they meet the criteria on day 1 of either conditioning chemotherapy (ASCT) or lymphodepleting chemotherapy (LDC) (CAR-T)
* Total bilirubin ≤ 1.5 x Institutional upper limit of normal (ULN) (except patients with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL), OR direct bilirubin ≤ ULN for patients with total bilirubin > 1.5 x ULN Patients must meet the parameter at screening if intended for ASCT or CAR-T treatment but have not yet received the cellular therapeutic. For patients enrolled after receiving ASCT or CAR T-cell therapy, patients will be eligible if they meet the criteria on day 1 of either conditioning chemotherapy (ASCT) or lymphodepleting chemotherapy (LDC) (CAR-T)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ 2.5 x institutional ULN Patients must meet the parameter at screening if intended for ASCT or CAR-T treatment but have not yet received the cellular therapeutic. For patients enrolled after receiving ASCT or CAR T-cell therapy, patients will be eligible if they meet the criteria on day 1 of either conditioning chemotherapy (ASCT) or lymphodepleting chemotherapy (LDC) (CAR-T)
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x institutional ULN Patients must meet the parameter at screening if intended for ASCT or CAR-T treatment but have not yet received the cellular therapeutic. For patients enrolled after receiving ASCT or CAR T-cell therapy, patients will be eligible if they meet the criteria on day 1 of either conditioning chemotherapy (ASCT) or lymphodepleting chemotherapy (LDC) (CAR-T)
* Creatinine clearance ≥ 30 mL/min estimated by the Cockcroft-Gault equation Patients must meet the parameter at screening if intended for ASCT or CAR-T treatment but have not yet received the cellular therapeutic. For patients enrolled after receiving ASCT or CAR T-cell therapy, patients will be eligible if they meet the criteria on day 1 of either conditioning chemotherapy (ASCT) or lymphodepleting chemotherapy (LDC) (CAR-T)
* International normalized ratio (INR) activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, unless participant is receiving anticoagulant therapy as long as INR or aPTT is within therapeutic range of intended use of anticoagulants Patients must meet the parameter at screening if intended for ASCT or CAR-T treatment but have not yet received the cellular therapeutic. For patients enrolled after receiving ASCT or CAR T-cell therapy, patients will be eligible if they meet the criteria on day 1 of either conditioning chemotherapy (ASCT) or lymphodepleting chemotherapy (LDC) (CAR-T)
* Patients with a known history of hepatitis C virus (HCV) infection who have undetectable HCV viral load at screening

  * Note: Patients must have completed curative anti-viral therapy at least 4 weeks prior to registration
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification

  * Note: To be eligible for this trial, patients should be class 2 or better
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Females of child-bearing potential (FOCBP) either practice complete abstinence or agree to use two reliable methods of contraception simultaneously. This includes ONE effective method of contraception and ONE additional effective contraceptive method. Women should use effective contraceptive methods beginning ≥ 28 days prior to initiating, study treatment, for the duration of study participation, and for at least 6 months following completion of therapy. As tazemetostat may interfere with hormonal contraception and render it ineffective, adequate contraception in this case would consist of a barrier method of birth control or abstinence.

Should a female patient become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Men treated or enrolled on this protocol must also agree to either practice complete abstinence or agree to use a latex or synthetic condom, even with a successful vasectomy (medically confirmed azoospermia), during sexual contact with a FOCBP from time of informed consent, for the duration of study participation (including during dose interruptions), and atleast 6 months after study drug discontinuation.

Male subjects must not donate semen or sperm from first dose of tazemetostat, during study treatment (including during dose interruptions), and for 6 months after discontinuation of study drugs.

NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy or bilateral salpingectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)

  * FOCBP must have a negative pregnancy test prior to registration on study
* Note: Serum or urine pregnancy test for females of childbearing potential. This should be performed within 28 days prior to registration. A pregnancy test will need to be repeated if cycle 1 day 1 is > 3 days after registration. Pregnancy test will also be done during maintenance phase with each cycle, for females of childbearing potential

Exclusion Criteria:

* Patients who are currently participating in or has participated in a study of an investigational agent or has used an investigational device within 28 days prior to the first dose of study intervention Exception: Out of spec CAR-T products are permitted
* Patients who have received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) or prior exposure to EZH2 inhibitors
* Patients who have received prior radiotherapy within 14 days of start of study intervention

  * Note: Patients must have recovered from all radiation-related toxicities, not require corticosteroids; patients with radiation pneumonitis are excluded
  * Note: A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Patients who have had major surgery within 4 weeks before the first planned dose of tazemetostat (i.e. cycle 2, day 1)

  * Note: Minor surgery (eg, minor biopsy of extracranial site, central venous catheter placement, shunt revision) is permitted within 3 weeks prior to the first planned dose of tazemetostat
* Patients with a known history of Human Immunodeficiency Virus (HIV) infection
* Patients with a known history of chronic hepatitis B (HBV) infection

  * Note: Patients who are hepatitis B surface antigen (HBsAg) positive, have received antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to registration are eligible. Patients should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention
* Patients with any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or myeloproliferative neoplasm (MPN)
* Patients with any prior history of T-cell lymphoblastic lymphoma (T-LBL)/ T cell acute lymphoblastic leukemia (T-ALL) or B cell acute lymphoblastic leukemia (B-ALL)
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab or tazemetostat
* Patients receiving medications or substances that are inhibitors or inducers of CYP450 enzymes are eligible as long as they meet the criteria
* Patients with a diagnosis of immunodeficiency or patients receiving chronic systemic glucocorticoids (in dosing exceeding 10 mg daily of prednisone equivalent) within 7 days prior to the first dose of study drug. Exceptions are:

  * To modulate symptoms of an adverse events (AE) that is suspected to have an immunologic etiology or related to prior CAR T-cell therapy
  * For the prevention of emesis
  * To premedicate for IV contrast allergies
  * To treat chronic obstructive pulmonary disease (COPD) exacerbations (only short-term oral or IV use in doses >10 mg/day prednisone equivalent)
  * For topical use or ocular use
  * Intraarticular joint use
  * For inhalation in the management of asthma or chronic obstructive pulmonary disease
* Patients who have active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs)

  * Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Patients who have received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention

  * Note: Administration of killed vaccines is allowed
* Patients who have a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease

  * Note: Patients with radiation pneumonitis are excluded
* Patients who have known additional malignancy that is progressing and/or receiving active therapy. Exceptions are patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin. Additionally carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are eligible
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following:

  * Hypertension that is not controlled on medication
  * Ongoing or active infection requiring systemic treatment
  * Active tuberculosis bacillus (TB) infection
  * History of allogenic tissue/solid organ transplant
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing

  * Note: Pregnant women are excluded from this study because pembrolizumab is a Class D agent with potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab, breastfeeding should be discontinued if the mother is treated with pembrolizumab and mother should abstain from breast feeding for 6 months. Tazemetostat should also not be used during pregnancy because there is potential risk for teratogenicity
* Patients with known active CNS metastases and/or carcinomatous meningitis
* Patients with severe hypersensitivity (≥ grade 3) to pembrolizumab and/or any of its excipients.
* Patients with presence of any clinically significant toxicities related to prior anticancer treatment (i.e., chemotherapy, immunotherapy, and/or radiotherapy), excluding transplant or CAR-T planned for current protocol, unless they have either resolved to grade 1 per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 OR are clinically stable and no longer clinically significant at the time the patient provides voluntary written informed
* Patients who have had an allogenic tissue/solid organ transplant
* Patients with the inability to take oral medication OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, vomiting) that might impair the bioavailability of tazemetostat
* Patients with a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2027-04-24 (Estimated); Study Completion 2028-11-24 (Estimated)

PRIMARY OUTCOMES:
Event free survival | At 6 months
  Event is defined as any of the following (whichever occurs first): death from any cause, progressive disease, failure to achieve complete or partial response by 6 months in CAR T patients, or start of new antineoplastic therapy due to efficacy concerns. Analysis will be performed using one sample exact test for proportions, comparing the 6-month EFS rate to the 45% historic control rate.

SECONDARY OUTCOMES:
Progression free survival | From autologous stem cell transplantation (ASCT) or chimeric antigen receptor (CAR) T-cell infusion until radiologically documented disease progression or death from any cause, whichever occurs first, up to 3 years
  Will be estimated using the method of Kaplan-Meier.
Overall survival | From ASCT or CAR T-cell infusion until death from any cause, up to 3 years
  Will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | From the start of CAR T or ASCT up to 30 days after treatment discontinuation
  Toxicity will be graded using the National Cancer institute Common Terminology Criteria for Adverse Events version 5.0.
Objective response rate (ORR) | At month 3, 6, 12, and 18
  ORR is defined as the proportion of patients achieving response of complete response (CR) or partial response (PR) at a specified time point. Will be reported as counts, proportions and the corresponding confidence intervals.
Complete response rate | At month 3, 6, 12, and 18
  CR rate is defined as the proportion of patients achieving a complete radiological response on positron emission tomography/computed tomography (PET/CT) (by Lugano criteria) from time of CAR T-cell infusion. Will be reported as counts, proportions and the corresponding confidence intervals.
Partial response rate | At month 3, 6, 12, and 18
  PR rate is defined as the proportion of patients achieving a partial radiological response on PET/CT (by Lugano criteria) from time of CAR T-cell infusion. Will be reported as counts, proportions and the corresponding confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Reem Karmali, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa